CLINICAL TRIAL: NCT01402245
Title: Comparison of Immune Response in Pneumococcal Pneumonia and After Vaccination
Brief Title: Targeting of Immune Response After Pneumococcal Vaccination
Acronym: PncHR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Anu Kantele, Helsinki UYniversity Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 411/E5/02; 383/E5/07 (Other: Ethics Committee, Dept. of Medicine, HUCH)
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2007-01

CONDITIONS: Pneumococcal Pneumonia
Keywords: pneumonia; pneumococcal polysaccharide vaccine; pneumococcal conjugate vaccine
MeSH Terms: conditions — Pneumonia, Pneumococcal; Pneumonia | interventions — Pneumococcal Vaccines; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pneumonia group (No Intervention): Patients with Pnc pneumonia
- PPV Group (Active Comparator): Volunteers immunized with Pnc polysaccharide vaccine
  Interventions: Biological: Pneumococcal polysaccharide vaccine
- PCV Group (Active Comparator): Volunteers immunized with Pnc conjugate vaccine
  Interventions: Biological: pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: Pneumococcal polysaccharide vaccine — Pneumococcal polysaccharide vaccine 0.5 ml i.m.
  Other Names: Pneumovax
  Arms: PPV Group
Biological: pneumococcal conjugate vaccine — pneumococcal conjugate vaccine 0.5 ml i.m.
  Other Names: Prevenar
  Arms: PCV Group

SUMMARY:
Pneumococcal polysaccharide vaccine does not confer protection against noninvasive pneumonia. The study aims to compare lymphocyte homing in pneumonia and in those receiving Pnc polysaccharide vaccine (PPV) or Pnc conjugate vaccine (PCV)

DETAILED DESCRIPTION:
Pneumococcal polysaccharide vaccine does not confer protection against noninvasive pneumonia. The study compares the homing profiles of Pnc-specific plasmablasts in 15 patients with pneumonia and in 15 volunteers receiving Pnc polysaccharide vaccine (PPV) and 12 volunteers receiving Pnc conjugate vaccine (PCV)

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 and <65 years of age.
* General good health.
* Written informed consent.
* No previous vaccination against Pnc
* No previous history of Pnc pneumonia
* In pneumonia: Diagnosis of Pnc pneumonia within a week

Exclusion Criteria:

* < 18 years, ≥65 of age.
* In vaccinees: Acute disease at the time of enrollment.
* Pregnancy or lactation.
* Known immunodeficiency or immune suppressive treatment.
* Any chronic illness that might interfere with the immune response
* Alcohol or drug abuse
* Any clinically significant history of known or suspected anaphylaxis or hypersensitivity (based on the investigator's judgement).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2005-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Expression of homing receptors on circulating plasmablasts in Pnc pneumonia and after vaccination | Day 0 and Day 7-10
  HR on circulating Pnc-specific plasmablasts are determined in patients with pneumonia on day 7-10, in vaccinees on days 0 and 7

CONTACTS AND LOCATIONS:
Overall Officials: Anu Kantele, MD PhD, Principal Investigator — Helsinki University Central Hospital
Locations (4):
- Finland (4):
  - University of Helsinki, Haartman institute, Dept. of Bacteriology and Immunology, Helsinki
  - Division of Infectious Diseases, HUCH, Helsinki
  - Division of Microbiology, HUSLAB, Helsinki University Central Hospital, Helsinki
  - University of Turku, Turku